CLINICAL TRIAL: NCT00747136
Title: A Prospective Evaluation of the WavSTAT® Optical Biopsy System to Target Esophageal Biopsies: An Adjunctive Tool to Assist the Endoscopist to Identify Dysplasia or Cancer
Brief Title: WavSTAT® Optical Biopsy System to Target Esophageal Biopsies
Status: Terminated | Type: Observational
Why Stopped: Study has been terminated for inadequate results
Sponsor: SpectraScience (Other)
Responsible Party: Sponsor
Other Study IDs: 010020-P-001
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's; Dysplasia; esophageal cancer; Patients
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — esophageal biopsies will be collected.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to demonstrate the clinical utility of the WavSTAT Optical Biopsy System as an adjunctive tool to improve the endoscopist's clinical sensitivity to identify dysplasia or cancer in the esophagus.

DETAILED DESCRIPTION:
In the clinical portion of this prospective study, the algorithm developed in the preclinical evaluation will be blindly tested using the pathologists' assessment of the biopsies as a gold standard to determine the clinical sensitivity and specificity of the WavSTAT Optical Biopsy System to identify dysplastic or cancerous tissue in the esophagus. In addition, the endoscopist's unaided clinical sensitivity and specificity to identify dysplasia or cancerous tissue will also be determined by recording the endoscopist's visual assessment of whether the physical biopsy has dysplasia or cancer or does not have dysplasia or cancer prior to performing the biopsy The endoscopist's assessment will be correlated and compared with the pathologist's interpretation. The clinical utility of the WavSTAT System to improve the endoscopist's clinical sensitivity to identify dysplasia or cancer in the esophagus will be evaluated by testing the hypothesis that the sensitivity of a WavSTAT-assisted endoscopic examination improves that of standard endoscopy alone.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 18 and 80 years of age.
* The patient is willing to sign an informed consent form.
* The patient is a candidate for endoscopic examination
* Female patients of child-bearing age, uncertain of pregnancy status, must have a negative pregnancy test.

Exclusion Criteria:

* The patient has congenital deformities, which preclude a physical biopsy procedure during endoscopy.
* The patient is pregnant or nursing by admission.
* The patient has other contraindications for physical biopsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Barrett's esophagus
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2008-08; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determine sensitivity/specificity to identify dysplasia/cancer in the esophagus WavSTAT System alone, endoscopist alone/combination of WavSTAT and endoscopist. Sensitivity of the endoscopist will be compared to combination of endoscopist and WavSTAT. | 9-15 months estimated

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Veterans Affairs, Kansas City, Missouri, United States